CLINICAL TRIAL: NCT04208438
Title: Non-Invasive Jugular Venous Blood Volume Assessment (BVI)
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: Mespere Lifesciences Inc. (Industry)
Responsible Party: Principal Investigator, Mark Favot, MD, Associate Professor of Emergency Medicine, Wayne State University
Other Study IDs: 20201216
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Ultrasound Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- BVI Cohort: Cohort to have ultrasound and Mespere BVI device applied.
  Interventions: Diagnostic Test: BVI Device; Diagnostic Test: Point-of-Care Ultrasound

INTERVENTIONS:
Diagnostic Test: BVI Device — Non-Invasive measurement of jugular blood volume using Mespere BVI device
Diagnostic Test: Point-of-Care Ultrasound — Point-of-Care ultrasound of external and internal jugular veins

SUMMARY:
The purpose of this study is to evaluate the ability of the Mespere Blood Volume Index (BVI) device to calculate the blood volume in the jugular veins by comparing the measurements from the device to volumetric measurements obtained with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater
2. English-speaking
3. No known medical conditions requiring treatment by a physician

Exclusion Criteria:

1. Substantial amount of neck hair preventing adhesion of the neck patch of the BVI
2. History of congenital heart disease
3. History of thoracic, neck or brain surgery
4. Inability to lay supine at 30 degrees incline or 60 degrees incline for the duration of the study measurements
5. Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Comparison of jugular vein blood volume | One Hour
  Comparison of measurement of blood volume in jugular vein using BVI and POCUS

SECONDARY OUTCOMES:
Comparison of changes in measurement of jugular venous blood volume | One Hour
  BVI vs POCUS at head of bed angle degrees 0, 30, and 60.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Biosciences Center - Clinical Research Service Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided